CLINICAL TRIAL: NCT02449590
Title: The Effects of Onion on Plasma Lipoproteins, Blood Pressure and Gene Expression in Overweight Humans - a Double-blinded, Randomized Cross-over Study
Brief Title: Onion, Cardiovascular Risk Markers and Gene Expression
Acronym: M197
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Lars Ove Dragsted (Other)
Collaborators: Instituto De Frio (Other Government); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Professor Lars Ove Dragsted, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M197
Record Dates: First submitted 2015-02-08; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Blood Pressure; Coagulation Delay
Keywords: Onion; Cardiovascular disease; metabolomics; Gene expression; Biomarker
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Onion powder (Active Comparator): Initial test meal contained 20g freeze dried onion powder in hot meals (1 potato soup and 1 meatball-meal daily). Subsequent daily meals contained 20g onion powder in the same meal formats.
  Interventions: Dietary Supplement: Onion powder
- Placebo (Placebo Comparator): Hot meals (1 potato soup and 1 meatball-meal daily)containing 8.5 g sucrose and 2 g soy protein instead of onion powder
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Onion powder — Hot meals with onion powder; 10 g/day onion powder corresponding to 100 g/day fresh onion in meals with potato and beef Intervention period 14 days.
  Arms: Onion powder
Dietary Supplement: Placebo — Hot meals without onion powder; Control meal with potato, beef, soy protein, and sucrose to match macronutrient composition of active treatment
  Arms: Placebo

SUMMARY:
AIMS:

The aims are to investigate whether:

* Increased intake of onion (powder) affects plasma lipid profile, blood pressure, indices of insulin sensitivity and blood coagulation.
* Increased intake of onion (powder) affects the expression/activity of enzymes in the defence against foreign substances, e.g. reactive oxygen species, and whether polymorphisms in some of the involved genes may modulate the effect.
* Polymorphisms involved in the metabolism/effect of bioactive components in onion modulate the excretion of metabolites or modulate some of the outcome variables in the study.

Other aims are to try to identify biomarkers for onion consumption in plasma, urine and feces and to investigate whether onion affects the secretion of fat and bile acids.

HYPOTHESES:

The investigators hypothesize that:

* 2 weeks of increased onion intake will improve the plasma lipid profile
* 2 weeks of increased onion intake will increase the metabolism of potentially harmful substances (such as ROS and free radicals) through a change in the expression or activity of certain enzymes.
* That these effects are modulated by common gene variants (polymorphisms)

DETAILED DESCRIPTION:
In a randomized controlled crossover design, participants will receive 2 daily meals with or without onion powder for 2 weeks. Between the two 2-week period is a 4-week wash-out period. One week before and during each intervention period, the participants will be instructed to avoid consumption of onion, garlic and all foodstuffs containing the same bioactive components (polyphenols, sulfur-molecules)as in onion. This includes a number of vegetables and fruits, condiments, tea, chocolate, red wine etc.

Fasting blood samples will be drawn before and after (on 2 separate days) each intervention period, where also weight and blood pressure are measured.

Participants will collect 24-hour urine and feces samples twice before and at completion of each intervention period.

After the fasting blood sampling on the first blood sampling day in each period, participants will receive a test meal (with 10 g onion powder or placebo, i.e. 8.5 g sucrose+ 2 g soy protein isolate). The acute effects will be studied by blood sampling and urine sampling 0, 2, 4 and 24 hours after the test meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI 25-40
* No daily medication (except thyroid hormone, stomach acid lowering drugs, mild blood pressure lowering drugs and anti-depressants)
* Not strenuous exercise >10 hours/week
* No blood donation 3 months before or during the study

Exclusion Criteria:

* Diabetes, CVD, hepatitis, HIV/AIDS
* Cancer or cancer treatment within last 6 months
* Smoking
* Simultaneous participation in other research projects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure from baseline to two weeks | baseline to two weeks
  Measured by a standard arm cuff by a trained bioanalyst

SECONDARY OUTCOMES:
Change in waist-to-hip circumference ratio | Change from baseline to two weeks
  Measured manually by a trained bioanalyst
Change in fecal microbiota profile | change from baseline to two weeks
  RFLP of 16S cDNA
Change in total cholesterol | change from baseline to 2, 4, and 24 hours and 2 weeks
  Total plasma cholesterol in lipoproteins measured by a clinical chemistry kit
Change in HDL cholesterol | change from baseline to 2, 4, and 24 hours and 2 weeks
  High density Lipoprotein Cholesterol in plasma measured by an immunokit
Change in plasma triacylglycerides | change from baseline to 2, 4, and 24 hours and 2 weeks
  Triacylglycerides in plasma measured by an immunokit
Change in blood coagulation parameters | 0-4 hours
  thromboelastography measurements, fibrinogen etc. in plasma
Change in whole-blood hematocrit | 0-14 days
  hematocrit by standard clinical chemistry
Change in whole-blood haemoglobin concentration | 0-14 days
  haemoglobin concentration by standard clinical chemistry
Change in body weight | 0-14 days
  Measured in triplicate on a calibrated balance
Change in serum VCAM-1 | 0-14 days
  Determined with standard kits
Change in serum IL-6 | 0-14 days
  Determined with standard kit
Change in serum TNF-alpha | 0-14 days
  Determined with standard kit
Change in faecal metabolic profiles | 0-14 days
  Untargeted metabolomics by LC-QTOF profiling of polar metabolites
Change in faecal pH | 0-14 days
  pH by a pH-meter in a 50% aqueous fecal slurry
Change in faecal bile acids | 0-14 days
  bile acids measured by LC-TQD
Change in urine metabolomic profiles | 0-14 days
  Untargeted metabolomics by LC-QTOF profiling of polar metabolites
Change in urine pH | 0-14 days
  pH by a pH-meter
Change in plasma insulin (multivariate ANOVA) | 0-14 days
  Insulin measured at baseline before meals and at 2, 4 and 24 hours, 2, 7 and 14 days after the start of intervention.
Change in plasma glucose (multivariate ANOVA) | 0-14 days
  Glucose measured at baseline before meals and at 2, 4 and 24 hours, 2, 7 and 14 days after the start of intervention.
Change in HOMA | 0-14 days
  Change in HOMA measured at baseline before meals and at 14 days after the start of intervention.
Change in ISI240 (Matsuda insulin sensitivity index 0-240) | 0-240 minutes
  Change in ISI240 measured from 0-240 minutes after the first test meal.
Change in erythrocyte Glutathione Reductase | 0-2 weeks
  Measured by automated colorimetric assays
Change in erythrocyte superoxide dismutase | 0-2 weeks
  Measured by automated colorimetric assays
Change in erythrocyte catalase | 0-2 weeks
  Measured by automated colorimetric assays
Change in erythrocyte glutathione peroxidase | 0-2 weeks
  Measured by automated colorimetric assays
Change in plasma untargeted metabolic profile | 0-2 weeks
  LC-QTOF profiling of polar metabolites and polar lipids
Change from baseline in leucocyte gene expression profile | 0, 2, 4 and 24 hours and 2 weeks
  Selected genes by RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — Dep Nutrition, Exercise and Sports, University of Copenhagen; Susanne G Bügel, PhD, Study Director — Dep Human Nutrition, LIFE, University of Copenhagen
Locations (2):
- Denmark (2):
  - Dep. Human Nutrition, LIFE, University of Copenhagen, Frederiksberg C
  - Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg C